CLINICAL TRIAL: NCT02299817
Title: Denosumab for Treating Periprosthetic Osteolysis After Uncemented Total Hip Arthroplasty A Randomized, Double-blind, Placebo-controlled Trial Using Volumetric Computed Tomography
Brief Title: Denosumab for Treating Periprosthetic Osteolysis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Olof Skoldenberg (Other)
Collaborators: Danderyd Hospital (Other)
Responsible Party: Sponsor-Investigator, Olof Skoldenberg, MD PhD, Danderyd Hospital
Organization: Danderyd Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EudraCT No: 2013-004940-48
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Osteolysis
MeSH Terms: conditions — Osteolysis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab (Active Comparator): Patients will receive a dose of 60 mg denosumab (1 ml solution) for a total of 6 doses with start on day one and every 6 months with last treatment at 30 months.
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Patients will receive a dose of placebo (1 ml solution) for a total of 6 doses with start on day one and every 6 months with last treatment at 30 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab — Prolia is used to treat osteoporosis (a disease that makes bones fragile) in women who have been through the menopause and in men who have an increased risk of fracture (broken bones). In women who have been through the menopause Prolia reduces the risk of fractures in the spine and elsewhere in the body, including in the hip.
  Prolia is also used to treat bone loss in men receiving treatment for prostate cancer that increases their risk of fracture. Prolia reduces the risk of fractures in the spine.
  Recently denosumab was found to be effective in preventing osteoporosis related fractures in post-menopausal women by blocking RANKL and thereby inhibiting the development and activity of osteoclast.
  Other Names: Prolia
  Arms: Denosumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objective is to study the efficacy of denosumab in reducing wear-induced osteolysis around uncemented acetabular implants used in total hip arthroplasty. Patients included in the study will receive the same dose of 60 mg denosumab or placebo (1 ml solution) for a total of 6 doses with start on day one and every 6 months with last treatment at 30 months. The primary endpoint will be the change in volume of the osteolytic lesion over 3 years measured (measured with 3D-CT in cm³).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85 years
* Short Portable Mental Status Questionnaire (SPMSQ) also named pfeiffers test ≥7
* Male and females
* The primary total hip arthroplasty performed between 7 to 20 years before inclusion.
* The primary total hip arthroplasty performed due to osteoarthritis or congenital dysplasia of the hip.
* Uncemented cup fixation
* Baseline osteolytic lesion of at least 4 cm³ and at most 40 cm³ around an uncemented acetabular component with a polyethylene liner.
* Participant is willing and able to follow study protocol and has provided informed consent prior to any study specific procedures.

Exclusion Criteria:

* For women of childbearing potential: Subject refuses to use 1 highly effective method of contraception (contraceptive pill, intra uterine contraceptive device) for the duration of the study and for 10 months after the last dose of study medication.
* For males with a partner of childbearing potential: Subject refuses to use a condom for the duration of the study and for 10 months after the last dose of study medication.
* For males with a partner who is pregnant: Subject refuses to use a condom for the duration of the study and for 10 months after the last dose of study medication.
* Pain in the operated hip (because the presence of hip pain in combination with an osteolytic lesion is an indication for revision surgery). VAS >3
* Previous revision surgery of the hip i.e. exchange of any inplant after the primary surgery
* Inflammatory arthritis
* Previous participation in clinical trials with denosumab or administration of commercial denosumab (Prolia™ or Xgeva™)
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s).
* Treatment with any intravenous bisphosphonate, fluoride (except for dental treatment) or strontium ranelate within 5 years prior to inclusion.
* Treatment with any oral bisphosphonate within 1 year prior to inclusion.
* Treatment with cortisol or cytostatic drugs within 6 months prior to inclusion.
* Administration of any of the following treatments 3 months prior to screening:

  * Anabolic steroids or testosterone
  * Glucocorticosteroids (≥ 5 mg prednisone equivalent per day for more than 10 days or a total cumulative dose of ≥ 50 mg)
  * Calcitonin
  * Calcitriol or vitamin D derivatives [vitamin D contained in supplements or multivitamins is allowed]
  * Other bone active drugs including anti convulsive (except benzodiazepines) and heparin
  * Chronic systemic ketoconazole, adrenocorticotrophic hormone, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, gonadotropin-releasing hormone agonists.
  * Androgen deprivation therapy
* Hypocalcaemia.
* Bone metabolic disorders (such as OI, PHPT, Paget)
* History of osteonecrosis of the jaw and/or recent tooth extraction or dental surgery; or planned invasive dental procedures during the study
* Serum 25-OH D <20 ng/ml
* Significant malabsorption including Celiac Disease, Short Bowel Syndrome, Crohn's Disease, Previous Gastric Bypass.
* Active cancer and/or malignancy in last 5 years (except cervical carcinoma in situ or basal cell carcinoma)
* History of solid organ or bone marrow transplant.
* Hypersensitivity to any components of study drug.
* Intolerance to calcium supplements.
* Pregnancy and/or currently lactating.
* Significantly impaired renal function as determined by a derived glomerular filtration rate (GFR) using Cockcroft Gault formula of 30 mL/min/1.73 m2
* Elevated transaminases ≥ 2.0 x upper limit of normal (ULN); Elevated total bilirubin (TBL) > 1.5 x ULN.
* Any condition or illness (acute, chronic, or history), which in the opinion of the Investigator might interfere with the evaluation of efficacy and safety during the study or may otherwise compromise the safety of the subject.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Volume of the osteolytic lesion | 3 years
  The change in volume of the osteolytic lesion over 3 years (measured with 3D-CT in cm³) is the primary endpoint variable: E〖fficacy〗_(3 years)=〖Volume〗_(3 years)-〖Volume〗_baseline.

SECONDARY OUTCOMES:
Volume of the osteolytic lesion | 2 years
  The change in volume of the osteolytic lesion over 2 years (measured with 3D-CT in cm³) 〖Efficacy〗_(2 years)=〖Volume〗_(2 years)-〖Volume〗_baseline.
Percentage change of the lesion over the study period | 3 years
  Percentage change of the lesion over the study period
Adverse events | 3 years
  Occurrence of AE´s

CONTACTS AND LOCATIONS:
Overall Officials: Olof Sköldenberg, MD, Ph.D, Study Director — Danderyds Hospital
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Axenhus M, Boden H, Kelly-Pettersson P, Skoldenberg O. Denosumab for treating periprosthetic osteolysis: a feasibility study. BMC Res Notes. 2025 Apr 8;18(1):151. doi: 10.1186/s13104-025-07216-0. PMID 40200363
- [Derived] Skoldenberg O, Rysinska A, Eisler T, Salemyr M, Boden H, Muren O. Denosumab for treating periprosthetic osteolysis; study protocol for a randomized, double-blind, placebo-controlled trial. BMC Musculoskelet Disord. 2016 Apr 23;17:174. doi: 10.1186/s12891-016-1036-5. PMID 27108405